CLINICAL TRIAL: NCT06932653
Title: SurgPASS: Reducing Deaths After Surgery in Low- and Middle-income Countries: A Pilot Cluster Randomised Trial
Brief Title: Reducing Deaths After Surgery in Low- and Middle-income Countries: A Pilot Cluster Randomised Trial
Acronym: SurgPASS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Lagos State University (Other); Christian Medical College and Hospital, Ludhiana (Unknown); University Teaching Hospital of Kigali (Unknown); Ministry of Health, Ghana (Other Government); Université d'Abomey-Calavi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SurgPASS
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Post-operative Complications
Keywords: pilot; cluster; surgical safety

STUDY DESIGN:
Intervention Model Description: Pilot cluster randomised trial.
Masking Description: Given this is a cluster trial, blinding of participants are not relevant as the entire cluster will be randomised to either the intervention or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Surgpass checklist and training champions (Experimental): A preoperative checklist for early recognition and treatment of acutely unwell surgical patients implemented through simulation training and clinical champions.
  Interventions: Other: SurgPASS - intervention
- Comparator - usual care (No Intervention): Usual care as per local practice at that site.

INTERVENTIONS:
Other: SurgPASS - intervention — SurgPASS consists of a preoperative surgical passport used for any patients requiring emergency laparotomy, a simulation training course and local clinical champions.
  Arms: Intervention - Surgpass checklist and training champions

SUMMARY:
SurgPASS is a pilot randomised cluster trial utilising a pre-operative checklist with the aim of reducing deaths after surgery. If SurgPASS is successful, the intervention will be implemented in a separate full-scale cluster randomised trial.

DETAILED DESCRIPTION:
Title: Reducing deaths after surgery in low- and middle-income countries: A pilot cluster randomised trial

Aim: This pilot randomised cluster trial aims to evaluate the feasibility of a large-scale cluster randomised trial to assess the effectiveness and implementation of a pre-operative checklist to reduce deaths after surgery. If this pilot study is successful, we aim to assess the intervention in a separate full-scale cluster randomised trial.

* Objective 1: To determine feasibility and fidelity of delivering the intervention.
* Objective 2: To determine the rate recruitment to inform how long it will take to recruit to a future cluster randomised trial.
* Objective 3: To obtain information on postoperative outcomes to help inform the outcomes used and sample size of the future cluster randomised trial.

Design: Pilot cluster randomised trial.

Inclusion: Adult (>18 years old) non-pregnant patients undergoing emergency abdominal surgery with an incision of ≥5cm.

Exclusion: Patients undergoing minimally invasive surgery, or surgery for appendicitis.

Intervention: SurgPASS is an intervention of a preoperative checklist for early recognition and treatment of acutely unwell surgical patients implemented through simulation training and clinical champions.

Comparator: Usual care as per local practice at that site.

Follow-up period: 30-days from surgery.

Number of participants: 300 participants: 25 participants in each of 12 clusters (hospitals), from 6 countries.

Outcomes: Since this is a pilot study, there are no pre-specified primary outcomes. However, there are four key outcomes of interest to assess ahead of the main phase randomised clinical trial.

* Outcome 1: Measure simulation training and checklist completion rate for participants undergoing surgery to refine future implementation (intervention clusters only)
* Outcome 2: Measure duration of time to recruit 25 participants per cluster (to determine duration of potential full trial)
* Outcome 3: Measure 30-day overall complication rates to inform overall sample size of potential full trial

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing emergency major abdominal surgery (i.e., midline or non-midline) with an incision greater than or equal to 5cm
* Patient must not be pregnant
* Adults only (greater than or equal to 18 years old)

Exclusion criteria:

* Minimally invasive surgery
* Surgery for appendicitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Training and checklist completion | Within 30 days postoperatively
  Measure simulation training and checklist completion rate for participants undergoing surgery to refine future implementation (intervention clusters only)

OTHER OUTCOMES:
Duration of time to recruit sample size per cluster | Within 6 months post cluster activation
  Measure duration of time to recruit 25 participants per cluster (to determine duration of potential full trial)
Complication rates | Within 30 days postoperatively
  Measure 30-day overall complication rates to inform overall sample size of potential full trial

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Principal Investigator — University of Birmingham
Locations (5):
- University of Abomey-Calavi, Abomey-Calavi, Cotonou, Benin
- Tamale Teaching Hospital, Tamale, Tamale, Ghana
- Christian Medical College (CMC) & Hospital, Ludhiana, Ludhiana, 141008, Ludhiana, India
- Lagos University Teaching Hospital (Hub), Lagos, Lagos, Nigeria
- University Teaching Hospital of Kigali (Hub), Kigali, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No
Hospital-level data will not be released or published. Country-level analyses will only be conducted with permission of lead investigators from each participating country. Local investigators may access their data across their country to perform country-level analyses (all participating hospitals should consent to their data being used in this way).